CLINICAL TRIAL: NCT03027960
Title: Empagliflozin in Heart Failure: Diuretic and Cardio-Renal Effects
Acronym: EMPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000020019
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure; Type II; Diabetes
Keywords: cardio-renal
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo, then empagliflozin (Experimental): Patients are randomized upon enrollment to determine whether they take empagliflozin or the matched placebo during the first 2-week treatment phase of the study. All patients then undergo a 2-week "washout period" before crossing over to the alternate therapy.
  Interventions: Drug: Empagliflozin; Drug: Placebo Oral Capsule
- Empagliflozin, then Placebo (Experimental): Patients are randomized upon enrollment to determine whether they take empagliflozin or the matched placebo during the first 2-week treatment phase of the study. All patients then undergo a 2-week "washout period" before crossing over to the alternate therapy.
  Interventions: Drug: Empagliflozin; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Empagliflozin — 10mg empagliflozin for a 2-week period
Drug: Placebo Oral Capsule — 10 mg placebo for a 2-week period

SUMMARY:
The investigators propose a small pilot proof of concept study to not only prove the existence of, but also probe the mechanisms underlying cardio-renal effects of empagliflozin in patients with heart failure. The investigators propose a 50 patient randomized, double-blind, placebo-controlled crossover study with patients with stable HF, type II diabetes and an eGFR >45ml/min/1.73 m2 who are chronically receiving loop diuretics.

DETAILED DESCRIPTION:
Study Objectives

1. Study the acute/short term effect and cardio-renal mechanisms of sodium-glucose cotransporter 2 (SGLT2) inhibition in patients with heart failure.
2. Determine the effect of chronic combined SLLGT2 and loop diuretic exposure in patients with heart failure.

Primary Outcomes

1. Aim 1 (Acute): Determine if acute SGLT2 inhibition will improve the natriuretic effect of a loop diuretic compared to placebo.
2. Aim 2 (Chronic): Determine the effect of 14 days of SGLT2 inhibition on blood volume.

ELIGIBILITY:
Inclusion Criteria:

* Stable HF as defined by:
* No hospitalization for >60 days
* Stable HF medications for >=2 weeks, and stable diuretics for 4 weeks
* Opinion of HF cardiologist that the patient is at their optimal volume status
* Chronic daily oral loop diuretic dose >=20mg furosemide equivalents
* Diagnosis of type II diabetes
* Patient monitors blood glucose regularly at home
* eGFR >=45 mL/min/1.73 m2
* >=18 years old

Exclusion Criteria:

* Active titration of chronic HF medications expected during the study period
* Use of a non-loop diuretic, aside from an aldosterone antagonist (<=25mg spironolactone or <=50mg eplerenone)
* Critical stenotic valvular disease, complex congenital heart disease, or prior heart transplant
* History of diabetic ketoacidosis, "brittle" diabetes, and/or frequent hypoglycemia or severe hypoglycemic episodes requiring emergent intervention (ER visit or EMS response, glucagon administration or forced oral carbs) in the last 6 months
* History of bladder dysfunction, incontinence, pyelonephritis, urosepsis, or frequent urinary tract infections
* Anemia (defined as hemoglobin <8g/dL)
* Pregnancy or breastfeeding
* History of serious hypersensitivity
* Participation in another trial with an investigational drug within the 30 days prior to informed consent
* Use of another SGLT-2 inhibitor
* Appears unlikely, or unable to participate in the required study procedures, as assessed by the study PI or research RN (ex: clinically-significant psychiatric, addictive, or neurological disease)
* Inability to give written informed consent or follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
urine sodium concentrations via ion selective electrodes | 36 days
  Determine if acute SGLT2 inhibition will improve the natriuretic effect of a loop diuretic compared to placebo.
  Measuring the natriuretic effect of a loop diuretic (placebo v acute SGLT2 inhibition) via urine sodium output.

SECONDARY OUTCOMES:
blood volume | 14 days
  Determine the effect of 14 days of SGLT2 inhibition on blood volume.
  Daxor Blood Volume Sample Collection
  1. Volumex Injection: The Volumex tracer (radiolabeled albumin) is injected as an intravenous bolus (IV-push). (As soon as the tracer injection begins, a stopwatch is started and never zeroed out. Running times are used for the entire procedure).
  2. Serial Blood Collection A series of 5 post-Volumex blood samples is collected, after tracer injection, allowing for complete mixing in the bloodstream.
  3. Sample Timing: Samples are ideally spaced ~6 minutes apart, and are collected approximately 12, 18, 24, 30 and 36 minutes after Volumex administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Testani, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao VS, Ivey-Miranda JB, Cox ZL, Moreno-Villagomez J, Maulion C, Bellumkonda L, Chang J, Field MP, Wiederin DR, Butler J, Collins SP, Turner JM, Wilson FP, Inzucchi SE, Wilcox CS, Ellison DH, Testani JM. Empagliflozin in Heart Failure: Regional Nephron Sodium Handling Effects. J Am Soc Nephrol. 2024 Feb 1;35(2):189-201. doi: 10.1681/ASN.0000000000000269. Epub 2023 Dec 11. PMID 38073038
- [Derived] Griffin M, Rao VS, Ivey-Miranda J, Fleming J, Mahoney D, Maulion C, Suda N, Siwakoti K, Ahmad T, Jacoby D, Riello R, Bellumkonda L, Cox Z, Collins S, Jeon S, Turner JM, Wilson FP, Butler J, Inzucchi SE, Testani JM. Empagliflozin in Heart Failure: Diuretic and Cardiorenal Effects. Circulation. 2020 Sep 15;142(11):1028-1039. doi: 10.1161/CIRCULATIONAHA.120.045691. Epub 2020 May 15. PMID 32410463